CLINICAL TRIAL: NCT03812276
Title: Prospective Observational Study of Neodent Implantable Devices of GM Line
Brief Title: Neodent Implantable Devices of GM Line
Status: Completed | Type: Observational
Sponsor: Neodent (Industry)
Responsible Party: Sponsor
Other Study IDs: CS.O.002
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Jaw, Edentulous; Jaw, Edentulous, Partially
Keywords: Dental Implants
MeSH Terms: conditions — Jaw, Edentulous; Jaw, Edentulous, Partially | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Study Group: Neodent Acqua GM Helix dental implants will be placed. Multiple implants may be placed in a single subject.
  Interventions: Device: Dental Implants

INTERVENTIONS:
Device: Dental Implants — Dental Implants will be used according to standard routine in daily practice, according to all indications as specified by the manufacturer in the IFU (informations for use).

SUMMARY:
Acqua GM (Grand Morse) Helix implants present an optimized implant design with adapted treatment protocol, allowing for treatment of patients with different bone qualities.

The objective of the study is to prospectively collect clinical data to confirm the long-term safety and clinical performance of Acqua GM Helix implants and GM prosthetic abutments in daily dental practice setting, by means of success and survival rates of these devices.

Devices will be used according to standard routine in daily practice, according to all indications as specified by the manufacturer in the IFU (instructions for use). patients will be followed for 36 months after implant placement.

DETAILED DESCRIPTION:
The study protocol was reviewed and approved by an Ethics Committee (CE) in Brazil.

The sample will be prospectively and consecutively selected and will consist of patients who are 18 years of age or older, who are in need of one or more dental implants and who qualify for placement of Neodent GM Helix implants. Informed consent in writing will be obtained from each patient participating in the study prior to any study related procedure.

Neodent Acqua GM Helix implants will be placed under local anesthesia and with adequate bone bed preparation, as recommended by the manufacturer. Multiple implants may be placed in a single subject. Implants will be placed 2mm below the alveolar ridge.

The selection of the prosthetic component and loading protocol (late or immediate) will be conducted according to the need of each subject and to the manufacturer's instructions (IFU). Thus, implant immediate loading may be performed (at the discretion of the surgeon) when primary stability reach at least 32 N.cm and the patient present physiological occlusion.

Data concerning the studied variables will be collected by fulfilling the Case Report Form (CRF), in the following stages: First visit (Screening); T0 - Implant(s) placement; TL - Implant loading; T6, T12, T24 and T36 - 6, 12, 24 and 36 months, respectively, after implant placement. A visit window of more or less one month is eligible for each of the planned intervals.

Standardized digital periapical radiographs, computed tomography scans and photographs will be obtained in an usual daily practice frequency, as determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Need of one or more dental implants;
* Qualify for placement of Neodent GM Helix implants.

Exclusion Criteria:

As exclusion criteria, solely the device contraindications according to the IFU (instructions for use) will be applied:

* Signs of allergy or hypersensitivity to the chemical ingredients of the material: titanium alloy;
* Presence of acute inflammatory or infectious processes in live tissue;
* Unsuitable bone volume or quality;
* Serious medical problems (e.g. bone metabolism disorders, blood clotting disorders, unsuitable healing capacity);
* Insufficient oral hygiene;
* Incomplete jawbone growth;
* Patient uncooperative and not motivated;
* Abuse of drugs or alcohol;
* Psychosis;
* Prolonged functional disorders which resist any treatment with medications;
* Xerostomia;
* Weakened immunological system;
* Diseases which require the use of steroids;
* Uncontrolled endocrinological diseases;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age or older who are in need of and who qualify for dental implant placement with GM Helix implants at the involved study centers. Patients that give written informed consent to participate in this clinical study.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-28 (Actual)

PRIMARY OUTCOMES:
Implant survival and success rates | 36 months after implant placement
  Implant survival will be defined as no loss of the implant at each follow-up. Evaluation of implant success will be assessed based on the criteria proposed by Buser et al. (1990).

SECONDARY OUTCOMES:
Implant survival and success rates | 6, 12 and 24 months after implant placement
  Implant survival will be defined as no loss of the implant at each follow-up. Evaluation of implant success will be assessed based on the criteria proposed by Buser et al. (1990).
Prosthetic survival and success rates | 12, 24 and 36 months after implant placement
  Prosthetic survival will be assessed as the prosthesis remaining in situ at each follow-up, irrespective of its condition. Success will be defined as the prosthesis that remained unchanged and did not require any intervention during the entire observational period.
Patient Satisfaction: OHIP-14 (Oral Health Impact Profile) questionnaire | 6, 12, 24 and 36 months after implant placement
  The Portuguese translation of OHIP-14 [18,19] questionnaire will be used to assess Oral Health Related Quality of Life (OHRQoL), as a measure of patient satisfaction with treatment. Scores will range from 0 (absence of negative impacts on oral health) to 28 (high frequency of negative impacts on oral health).
Clinician Satisfaction: VAS (Visual Analogue Scale) questionnaire | Implant placement, 12, 24 and 36 months after implant placement
  The assessment will be performed by means of a questionnaire using a visual analog scale (VAS) in the form of a 10 cm horizontal line, where 0 (left end) indicates minimum satisfaction and 10 (right end) indicates maximum satisfaction. The clinician will be instructed to mark the position considered to best represent their degree of general satisfaction with patient treatment. The score will be measured in centimeters from the left end of the line to the marked point.
Rate of adverse events related to the implant, prosthesis, surgery and oral health | Implant placement, 6, 12, 24 and 36 months after implant placement
  Determined by inquiring with the patient and clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Larissa Trojan, PhD, Study Chair — Neodent
Locations (2):
- Brazil (2):
  - Instituto Latino Americano de Pesquisa e Ensino Odontológico (ILAPEO), Curitiba, Paraná
  - Universidade Positivo, Curitiba, Paraná

IPD SHARING:
Plan to Share IPD: No